CLINICAL TRIAL: NCT03214575
Title: Ultrasound Guided Central Venous Vascular Access - Novel Needle Navigation Technology Compared With Conventional Method: A Prospective Randomized Study
Brief Title: Ultrasound Guided Central Venous Vascular Access - Novel Needle Navigation Technology Compared With Conventional Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Mohd Shahnaz, MBBS, M Anes, Assoc. Prof., University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-16-334-29476
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Critically Ill
Keywords: Central Venous Vascular Access; Intensive Care Unit; Needle Navigation Technology
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional method (Active Comparator): For the Conventional method of ultrasound guided central venous catheter insertion,we use the ultrasound machine, eZono 4000 and linear array transducer L3-12NGS (3-12 MHz)
  Interventions: Device: Conventional method
- GPS method (Experimental): For the GPS method, we use the ultrasound machine, eZono 4000 with built-in adaptive needle recognition software called eZGuide (eZono, Jena, Germany) and linear array transducer L3-12NGS (3-12 MHz).
  Interventions: Procedure: GPS Method

INTERVENTIONS:
Device: Conventional method
  Arms: Conventional method
Procedure: GPS Method
  Arms: GPS method

SUMMARY:
Background: Central venous catheter (CVC) insertion is a very common procedure in the intensive care setting. A recent international guidelines advocated the use of ultrasound for routine internal jugular CVC insertion. The needle navigation technology is a new innovation, also known as guided positioning system (GPS) which allows clinician to visualize the needle position and trajectory in real time as it approaches the target. We hypothesised that the use of GPS would increase success rate and decrease performance time in vascular access procedures.

Objectives: To compare the success, efficacy and safety of the procedure using the ultrasound guidance (UG) with conventional versus GPS method.

Methods: This was a prospective randomized controlled study in a single centre - intensive care unit. 100 patients were randomized into two groups (50 each each). Subjects would receive CVC insertion via internal jugular vein using ultrasound guidance out of plane approach by conventional versus GPS method. Outcomes measured were the procedure efficacy, safety, level of operators' experience and their satisfaction.

DETAILED DESCRIPTION:
Introduction Central venous catheter (CVC) insertion is a very common procedure in the intensive care setting. A recent international guideline advocates the use of ultrasound for routine internal jugular central venous catheter insertion1. The needle navigation technology is a new innovation, also known as guided positioning system (GPS) which allows clinician to visualize the needle position and trajectory in real time as it approaches the target. We hypothesised that the use of GPS would increase success rate and decrease performance time in vascular access procedures. The objectives of this study are to compare the success, efficacy and safety of central venous catheter insertion via internal jugular vein using the ultrasound guidance with conventional method versus needle navigation technology.

Methods:

This was a prospective randomized controlled study. It was conducted in a single centre - intensive care unit (ICU), University of Malaya Medical Centre, Kuala Lumpur, Malaysia from February 2016 to October 2016. The ethic committee approval was obtained from the Malaysian medical research and ethics committee, MREC at the www.nih.gov.my (NMRR-16-334-29476).

The inclusion criterion was patients in the ICU who required central venous vascular access. The exclusion criteria were refusal to participate in this study by patient or their legal representative and patient with known history of difficult central venous access at internal jugular vein (IJV). The procedure operators were doctors in anaesthesia residency program with various level of experiences classified into 3 groups: 1 to < 2 years, 2 to < 3years, 3 years and above. Simply speaking all the operators have had previous training in ultrasound guided vascular access procedure. This would ensure that patient's safety is not compromised.

Study would be proceeded after obtaining consent from patient or the next of kin. The emergency verbal consent would be taken if the next of kin was not immediately available with subsequent written consent to follow. The available operator would perform CVC insertion via IJV using ultrasound guidance out of plane approach either with conventional method or needle guidance technology.

Study Protocol:

After obtaining consent, a computer generated randomisation would be assigned to either using the conventional or GPS method. Identified operators using GPS method would receive a standard 5 minute briefing on the needle guidance technology and got to practice with the new technology using the vascular phantom (Blue Phantom Inc., Bothell, WA, USA). The operators were allowed to practice until they were ready to perform on real patient.

All procedure would be performed using the ultrasound machine, eZono 4000 with eZGuide (eZono, Jena, Germany) and linear array transducer L3-12NGS (3-12 MHz). This ultrasound machine2 has a built-in adaptive needle recognition software called eZGuide. The navigation technology of the ultrasound device is based on an electromagnetic field that communicates with a transducer and an electromagnetic sensor sheathed by a vascular access needle. Needle movements and related magnetic field variation allow navigation system to compute the locations of the transducer and needle in the three dimensional space. The ultrasound screen would display colour coded alignment of the needle and the position of the tip relative to the imaging plane (Figure 1). Superimposed on the image is the real-time electronic needle guidance system. The dashed line represents the predicted needle trajectory. The red box represents the depth that the needle will cross the plane of the ultrasound. The solid lines on either side of the dashed line represent the actual depth of the needle. The top left corner shows a diagram of the transducer-needle relation. This allowed the user to identify the correct needle trajectory, prior to puncturing the patient's skin and maintain the chosen route to the target anatomy. Operators assigned to use GPS method would have activated the eZGuide software while those performing conventionally would have the software technology turned off when using the ultrasound machine.

The procedure time was measured in seconds using a stopwatch. The performance time was defined as time measured from placing the needle on the skin to successful vessel puncture as indicated by blood withdrawn into the syringe.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the ICU who required central venous vascular access.

Exclusion Criteria:

* Refusal to participate in this study by patient or their legal representative and patient with known history of difficult central venous access at internal jugular vein (IJV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
The procedure efficacy justified by successful cannulation. | 0-120 seconds
  The procedure efficacy justified by successful cannulation based on the performance time and number of attempts,

SECONDARY OUTCOMES:
Safety of procedure and complications. | During and within 24 hours after procedure.
  The safety of the procedure by identifying any potential complications occur, i.e. secondary tissue injury, hematoma, bleeding, pneumothorax, haemothorax or arterial puncture.
Operators' satisfaction. | within 1 week
  Level of operators' satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mohd Shahnaz Hasan, MBBS, Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: Undecided